CLINICAL TRIAL: NCT00619723
Title: A 12-week, Randomized, Double-blind, Parallel-group, Placebo-controlled Trial of Citicoline as an add-on Therapy Will be Conducted in 200 Outpatients With Bipolar I Disorder and Cocaine Dependence.
Brief Title: Citicoline for Bipolar 1 Disorder and Cocaine Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sherwood Brown, E. Sherwood Brown, M.D., PhD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 122007-039; 1R01DA022460-01A2 (NIH)
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Bipolar Disorder; Cocaine Dependence
MeSH Terms: conditions — Bipolar Disorder; Cocaine-Related Disorders | interventions — Cytidine Diphosphate Choline; Sugars; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citicoline (Active Comparator): Participants will receive active medication throughout the study. Citicoline will be given beginning at two capsules (500 mg/day) with an increase to four capsules (1000 mg/day) at week 2, six capsules (1500 mg/day) at week 4, and eight capsules (2000 mg/day) at week 6. Doses will be decreased, based on clinician judgment, due to side effects.
  Interventions: Drug: Citicoline; Behavioral: Cognitive Behavioral Therapy (CBT)
- Placebo (Placebo Comparator): Participants will receive placebo identical in appearance to Citicoline throughout the study. Placebo will be given beginning at two capsules (500 mg/day) with an increase to four capsules (1000 mg/day) at week 2, six capsules (1500 mg/day) at week 4, and eight capsules (2000 mg/day) at week 6. Doses will be decreased, based on clinician judgment, due to side effects.
  Interventions: Drug: Placebo; Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: Citicoline — Citicoline is a psychostimulant/nootropic. It is an intermediate in the generation of phosphatidylcholine from choline.
  Other Names: Cytidine diphosphate-choline (CDP-Choline); Cytidine 5'-diphosphocholine
  Arms: Citicoline
Drug: Placebo — Inactive ingredient matching the active medication in appearance.
  Other Names: Sugar pill
  Arms: Placebo
Behavioral: Cognitive Behavioral Therapy (CBT) — Participants will receive manual-driven Cognitive Behavioral Therapy (CBT: two sessions each week for 4 weeks followed by weekly sessions, total 16 sessions) specifically designed for persons with bipolar 1 disorder and substance abuse, and provided by a therapist with experience in CBT.

SUMMARY:
A 12-week, randomized, double-blind, parallel-group, placebo-controlled trial of citicoline as an add-on therapy will be conducted in 200 outpatients with bipolar I disorder and cocaine dependence. Patients will complete mood and memory assessments weekly, in addition to completing self-report measures for cocaine (and other substances, like alcohol) use and craving. Participants will receive manual-driven Cognitive Behavioral Therapy (CBT: two sessions each week for 4 weeks followed by weekly sessions, total 16 sessions) specifically designed for persons with bipolar 1 disorder and substance abuse, and provided by a therapist with experience in CBT. The sessions may be videotaped for training purposes and may be viewed by the researchers, the therapist, and Dr. Schmitz, a clinical researcher at the University of Texas Houston who is the developer of the CBT for bipolar disorder and substance dependence used in the study. Before being videotaped, the patient will sign an "Authorization for Audio Recordings, Photography, or Other Images for Non-Treatment Purposes" to further understand how the videotape will be used, and by whom. The patient will be given the option to review their videotape to view their therapy session. Once the patient has completed all study procedures, or had discontinued the study, the tape will be destroyed, until then the tape will kept in the patient's confidential study file. Further, patients will return to the clinic three times a week for urine drug tests (UDS). 200 patients are expected to be consented for this study and all study procedures will take place at the clinic on the University of Texas Southwestern Medical Center campus.

All non-study medications are not part of the study. Non-study medication will be verbally self-reported by the patient at the time of enrollment into the study. The patient will be responsible for the costs of their non-study related medications. The patient will manage their non-study medications with their personal doctor, including any changes in these medications. However the protocol has concomitant medication algorithm in the event that a change in the medication schedule needs to be made by a study doctor. If a study doctor requests a laboratory test for the patient, it will be paid for by the clinic. Otherwise, the patient will be responsible for all costs (including laboratories) associated with their non-study medications.

DETAILED DESCRIPTION:
There will be 13 study visits where patients complete assessments, urine drug screen, and cognitive behavioral therapy (CBT). Patients will need to come to the clinic two more times in the same week to complete additional urine drug screens, for a total of 26 visits dedicated to drug screens. In the first four weeks of the study, the patients will need complete cognitive behavioral therapy twice a week, so they will need to return to the clinic for an additional visit during their first month of participation in the study. These additional visits for CBT can be combined with the urine drug screen visits, for a maximum of 39 study visits to be completed.

At the first study visit (baseline), informed consent will be obtained including a review of inclusion and exclusion criteria. A Structured Clinical Interview (SCID) Clinician Version will be performed by a research assistant to establish the diagnoses of bipolar I disorder and cocaine dependence and establish concurrent comorbid illnesses. In addition, a psychiatrist with extensive experience working with patients with bipolar 1 disorder and substance abuse will confirm diagnoses based on a clinical evaluation.

During the baseline visit, eligible participants will then be given the Inventory of Depressive Symptomatology-Self Report 30-item version (IDS-SR30), Hamilton Rating Scale for Depression 17-item version (HRSD17), Young Mania Rating Scale (YMRS), Cocaine Craving Questionnaire 45-item weekly version (CCQ), Addiction Severity Index (ASI), Psychobiology of Recovery in Depression III Somatic Symptom Scale (PRD-III), a neurocognitive battery, and a urine drug screen (UDS). The battery of neurocognitive assessments will be repeated at weeks 3, 6, and 12 (exit).

During the same visit, cocaine use in the past week (dollar amount spent/week and days used/week) will be assessed by patient self-report. Use of and craving for other substances (benzodiazepines, barbiturates, alcohol, opiates, phencyclidine, and cannabis) will also be assessed by self-report of dollar amount and days used in the past week, UDSs, and with 100-mm single item visual analog craving scales. Craving for other substances will be measured using the Clinical Institute Withdrawal Assessment of Alcohol Use-Revised (CIWA-AR), Clinical Opiate Withdrawal Scale (COWs) and Benzodiazepine Withdrawal Symptom Questionnaire (BWSQ).

Medical and psychiatric histories will also be obtained at the baseline visit. Blood will be drawn for routine laboratory analyses including a complete blood count (CBC) and Sequential Multiple Analysis (SMA-20) at baseline and exit. The SMA-20 is a chemical test performed on serum (the portion of blood without cells). These tests include total cholesterol, total protein, various electrolytes (including sodium, potassium, chlorine), and chemicals that help the liver and kidney breakdown various substances. Both times we will draw approximately 2 tablespoons of blood, for a total of four tablespoons drawn over the course of the study.

A physical examination will be performed at baseline and exit. Women of childbearing potential will receive a urine pregnancy test and will be counseled about effective contraceptive methods. The pregnancy test will be repeated at week 4, 8, and 12 (exit) visits. The baseline visit will last approximately 3.5 hours; subsequent weekly visits will last approximately an hour.

A psychiatrist will assess the participants at baseline and weekly follow-up visits and will participate in the informed consent process. At each weekly assessment the HRSD17, IDS-SR30, YMRS, CCQ, and assessment of drug use in the past week will again be evaluated and a urine sample obtained. Adherence with study medication will be assessed through the use of the Medication Event Monitoring System (MEMS) metered dosing caps (primary measure) and pill counts.

Participants will return once each week for assessments, with additional visits for UDSs. Three UDSs will be obtained each week (Monday-Wednesday-Friday). UDS visits should last approximately 15 minutes.

The ASI will be repeated every 4 weeks. In addition, all participants will receive manual-driven CBT (two sessions each week for 4 weeks followed by weekly sessions, total 16 sessions) specifically designed for persons with bipolar 1 disorder and substance abuse, and provided by a therapist with experience in CBT. Each CBT session will last approximately one hour.

Citicoline or placebo will be given orally beginning at 500 mg/day (two tablets) with an increase to 1000 mg/day (four tablets) at week 2, 1500 mg/day (six tablets) at week 4, and 2000 mg/day (eight tablets) at week 6. Doses will be decreased if needed due to side effects.

After completing the study, patients will, if necessary, be provided standard care for bipolar 1 disorder, including continued care until symptom stabilization and referral to an outside clinic can be arranged. This post-study treatment will be provided by a blinded psychiatrist to maintain the integrity of the blind. We will make a strong effort, through phone calls and letters, to make contact with participants who withdraw from the study prior to completion to encourage them to return for a final assessment and to obtain information on the reasons for stopping treatment, perceptions of the research study and medication, and to help with arrangements for further treatment for their psychiatric illnesses outside of the study.

ELIGIBILITY:
Criteria for Inclusion of Subjects:

* Outpatients with a diagnosis of bipolar I disorder on the SCID and confirmed by interview with PI or co-I.
* Current diagnosis of cocaine dependence, cocaine use (by self-report) within 7 days prior to baseline, and a cocaine-positive urine at baseline
* Current mood state of depressed or mixed (depression plus mania) based on SCID interview using Diagnostic and Statistical Manual (DSM-IV) criteria.
* Baseline HRSD17 score < 35 and YMRS score < 35.
* On a stable medication regimen that may include mood stabilizers, antidepressants or other psychotropic medications (e.g. lithium, divalproex/valproic acid) for at least 14 days.
* Age 18-65 years old.
* Men and women.
* English speaking individual, who can also read English. The neurocognitive measures used in this study are not available in any other languages, and must be read by the patient. There is no ability to collect this data in another manner; therefore people unable to read English may not be enrolled for participation in this study.

Criteria for Exclusion of Subjects:

* Bipolar disorders other than bipolar I (e.g., bipolar II, not otherwise specified (NOS), or cyclothymic disorders) based on the SCID and confirmed through clinical assessment by PI or co-I.
* Mental retardation or other severe cognitive impairment, prison or jail inmates, pregnant or nursing women, or women of childbearing age who will not use hormonal contraceptives, abstinence, or other acceptable methods of birth control during the study.
* Currently experiencing psychotic features (delusions, hallucinations, disorganized thought processes).
* Initiation of antidepressants, mood stabilizers, or psychotherapy within the past 14 days.
* High risk for suicide, defined as any suicide attempt in the past 6 months, or current suicidal ideation with plan and intent or a score of ≥ 2 on the suicide item of the HRSD17.
* Intensive outpatient treatment for substance abuse (however, Alcoholics Anonymous (AA), Narcotics Anonymous (NA) meetings, or weekly therapy/counseling for bipolar disorder or substance use for at least 28 days prior to randomization will be encouraged).
* Severe or life-threatening medical condition (e.g., hepatic cirrhosis, congestive heart failure, terminal cancer), laboratory or physical examination findings consistent with serious medical illness (e.g., severe edema, atrial fibrillation, dangerously abnormal electrolytes), history of severe alcohol withdrawal in the past (e.g., delirium tremens), or current clinically significant alcohol (Clinical Institute Withdrawal Assessment for Alcohol Scale [CIWA-AR] score > 8 at baseline), opiate (Clinical Opiate Withdrawal Scale [COWS] score > 4 are baseline) or sedative/hypnotic/anxiolytic (Benzodiazepine Withdrawal Symptom Questionnaire [BWSQ] > 2).
* Drug of choice is not cocaine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, MD, PhD, Principal Investigator — UTSouthwestern Medical Center at Dallas
Locations (1):
- Exchange Park Center, American General Building (Bass)- PNE: FL8, STE 828, Dallas, Texas, United States

REFERENCES:
- [Derived] Brown ES, Todd JP, Hu LT, Schmitz JM, Carmody TJ, Nakamura A, Sunderajan P, Rush AJ, Adinoff B, Bret ME, Holmes T, Lo A. A Randomized, Double-Blind, Placebo-Controlled Trial of Citicoline for Cocaine Dependence in Bipolar I Disorder. Am J Psychiatry. 2015 Oct;172(10):1014-21. doi: 10.1176/appi.ajp.2015.14070857. Epub 2015 May 22. PMID 25998279

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Citicoline | Placebo
Started | 63 | 67
Completed | 61 | 61
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citicoline | Placebo | Total
Number analyzed (Participants) | 63 | 67 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 67 | 130
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (9.1) | 43.6 (8.3) | 42.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 27 | 43
  Male | 47 | 40 | 87
Region of Enrollment [Number; unit: participants]
  United States | 63 | 67 | 130

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Presence of a Cocaine-Positive Urine Screen
Description: Cocaine use frequency was measured by the presence or absence of a cocaine-positive urine screen. Drug screens were obtained thrice-weekly for 12 weeks. All participants who completed the baseline assessment and at least one additional assessment were included in the primary analysis. Missing data were imputed as cocaine positive.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 61 | 61
percentage of participants | 59.0 | 49.2

2. Secondary Outcome: Depressive Symptoms Measured Using the Hamilton Rating Scale for Depression (HRSD)
Description: As part of HRSD, the patient is rated by a clinician on 17 items that measure depressive symptom severity. The total score is calculated by summing the responses across all items. Lower scores (closer to 0) indicate the absence of depressive symptoms, while higher scores indicate the presence of depressive symptoms. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2 (0 = not present; 2 = severe). The scale range of scores is 0-52.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 61 | 61
units on a scale | 17.9 (5.6) | 18.0 (6.3)

3. Secondary Outcome: Manic Symptoms Measured Using Young Mania Rating Scale (YMRS)
Description: The Young Mania Rating Scale (YMRS) is a clinician-rated scale that has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. The total score is calculated by summing answers to all the item on the scale, with a higher score indicative of more severe mania symptoms. The scale total score ranges from 0 (absence of manic symptoms) to 60 (severe manic symptoms).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citicoline | Placebo
Number analyzed (Participants) | 61 | 61
units on a scale | 10.2 (5.9) | 10.1 (6.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study between 2008 and 2012. Each participant was enrolled for 12 weeks. Adverse events were collected for the full 12 weeks, beginning after consent was signed.
Description: Adverse events were assessed by a weekly questionnaire at each appointment.
Arm/Group | Citicoline | Placebo
Serious Adverse Events (participants affected / at risk) | 5/61 | 8/61
Other Adverse Events (participants affected / at risk) | 1/61 | 4/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Citicoline (N=61) | Placebo (N=61)
Overnight hospitalization due to motor vehicle accident (Musculoskeletal and connective tissue disorders) | 0 | 1 — Released from hospital with severe bruising only. Deemed as a serious, unexpected and non-study related adverse event.
Inpatient hospitalization due to improperly healing bones from previous accident (Musculoskeletal and connective tissue disorders) | 1 | 0 — Event deemed as serious, unexpected and non-study related.
Abnormal EKG indicating previous heart damage (Cardiac disorders) | 0 | 1 — Subject reported after receiving abnormal EKG on 2/18/10, that he had experienced chest pains after cocaine use in January (was not reported to study personnel at time). Blind was broken and subject sent to ER for workup.
Rape (Reproductive system and breast disorders) | 1 | 0 — Subject informed staff that she was raped. Subject denied physical injuries and was encouraged by study doctor to follow-up with primary care physician. Deemed serious, unexpected, and non-related to study medication.
Suicidal Ideation (Psychiatric disorders) | 0 | 1 — Subject reported suicidal ideation during study visit. Subject was assessed by study doctor and asked to agree to hospitalization. Subject refused and ran from office. Subject was contacted next day was deemed stable but withdrawn from study.
Hospitalization due to subacute pulmonary embolism (Cardiac disorders) | 0 | 1 — Subject hospitalized for 4 days due to subacute pulmonary embolism and was there treated with Coumadin. Subject withdrawn from study and encouraged to follow-up with physician. Event deem serious, expected, and unrelated to study medication.
Labs results indicating Leukopenia and Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 — Subjects baseline blood lab results indicated abnormal white blood cell and platelet count. Labs were repeated and revealed similar result. Subject was withdrawn from study. Event deemed as serious, unexpected and unrelated to study medication.
Suicidal Ideation (Psychiatric disorders) | 0 | 1 — Ideation reported during study visit. Subject assessed by study personnel and created safety plan. Subject reported later in the day that ideation worsened and voluntarily committed himself to hospital. Serious, expected, unrelated to study.
Ankle injury (Musculoskeletal and connective tissue disorders) | 0 | 1 — Subject experienced an ankle injury while mowing the lawn. Subject was assessed at the ER and given pain medication. Adverse event deemed as serious, unexpected, and unrelated to study medication.
Alcohol poisoning (General disorders) | 0 | 1 — Subject reported to ER due to nausea, vomiting, faintness following drinking binge. At ER, subject deemed to have alcohol poisoning and given IV fluids and released same day. Event deemed to be serious, unexpected, and unrelated to study medication.
Hairline fracture due to car accident (Musculoskeletal and connective tissue disorders) | 1 | 0 — Subject reported to ER after car accident. Hospitalized overnight and diagnosed with hairline fracture in ribs. Event deemed as serious, unexpected, and not related to study medication.
Hospitalization due to flu-like symptoms (General disorders) | 1 | 0 — Subject hospitalized for 2 days due to flu-like symptoms. All tests at hospital came back negative and subject was released. Event deemed as serious, unexpected and unrelated to study medication.
Hospitalization due to pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Subject hospitalized for 5 days due to flu-like symptoms. In ER, subject diagnosed with pneumonia and treated with IV fluids and medication. Event deemed as serious, unexpected and unrelated to the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Citicoline (N=61) | Placebo (N=61)
ER visit due to bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Subject went to ER due to bronchitis and was given antibiotics and released the same day.
Superficial cuts and bruising due to attack (General disorders) | 0 | 1 — Subject reported being attacked by a man with a knife while returning home from work. Subject had two 1-inch superficial cuts on right hip and minor bruise to left upper chest. Event deemed non-serious, unexpected and non-study related.
Lacerations on face due to fall (Skin and subcutaneous tissue disorders) | 0 | 1 — Subject reported slipping on water resulting in a fall on a glass vase, which led to multiple lacerations on face. Subject received stiches at ER and medication and sent home same day. Event deemed non-serious, unexpected and not related to study.
ER visit for breathing treatment (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Subject reported visiting ER for asthma breathing treatment. Subject not admitted to hospital and left after receiving breathing treatment. Event deemed non-serious, expected, and non-study related.
ER visit after slicing head on razor wire (Skin and subcutaneous tissue disorders) | 0 | 1 — Subject received 9 staples in ER and released same day. Event deemed as non-serious, unexpected and non-study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No